CLINICAL TRIAL: NCT00565773
Title: Use of Belatacept During Post Depletional Repopulation to Facilitate Tolerance in Renal Allograft Recipients
Brief Title: Belatacept Post Depletional Repopulation to Facilitate Tolerance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allan D Kirk, MD, PhD (Other)
Collaborators: Bristol-Myers Squibb (Industry); Duke University (Other)
Responsible Party: Sponsor-Investigator, Allan D Kirk, MD, PhD, Professor, Emory University
Organization: Emory University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00005064; Grant # FD-R-003539 (Other Grant/Funding Number: FDA Office of Orphan Products); BMS IM103-036 (Other: Other)
Record Dates: First submitted 2007-11-28; First posted 2007-11-30 (Estimated); Results first posted 2020-01-30 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Organ Transplantation
MeSH Terms: interventions — Abatacept; Sirolimus; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Immunosuppressive medications (Experimental): Renal transplant recipients will be given an experimental combination of immunosuppressive drugs. Participants will receive a single dose of alemtuzumab on the day of transplantation and will receive belatacept and sirolimus for 1 year.
  At the time of transplant, all patients will receive a single dose of 500 mg of methylprednisolone IV over 30 minutes, followed within 1 hour by an IV infusion of 30 mg of alemtuzumab over 3 hours.
  Interventions: Drug: Belatacept; Drug: Sirolimus; Drug: Alemtuzumab

INTERVENTIONS:
Drug: Belatacept — Belatacept will be given within 24 hours of transplantation via a peripheral intravenous catheter at a dose of 10mg/kg (actual body weight) infused over 30 mins. The dose will be repeated on study days 4 (post op day 3) and 8 (post op day 7), then every 2 weeks for 5 additional doses. Thereafter, belatacept will be given once every 4 weeks (+/- 3 days) at 10mg/kg through 6 months then at 5mg/kg indefinitely.
  Other Names: LEA29Y; Nulojix
Drug: Sirolimus — Sirolimus will be started on postoperative day 1 at a dose of 2 mg per day orally. Doses will be adjusted to maintain 24-hour trough levels of 8-10ng/ml until the drug is weaned. Toxicity attributable to sirolimus (e.g., mouth ulcers, arthralgias) will prompt dose reduction to address clinical concerns in this regard. If sirolimus trough levels need to be reduced below 4ng/ml to control drug side effects, the patient will be considered intolerant to the drug and will be changed to other medications.
  Other Names: Rapamycin
Drug: Alemtuzumab — All participants will receive a single dose of 30 mgs of alemtuzumab on the day of transplantation.
  Other Names: Campath; Lemtrada

SUMMARY:
Acute rejection is a common problem after a kidney transplant. Rejection can occur when the kidney recipient's immune system tries to attack (or reject) the new kidney. Rejection typically most often develops in the first few months after a transplant.

This single center study will seek to determine if a new combination of anti-rejection medications, including the recently FDA approved drug called Belatacept, is better than the current standard anti-rejection drug regimen at preventing rejection. Also to be determined will be whether the new combination of drugs will allow participants to wean off their oral anti-rejection medications over time.

This study will test the safety and effectiveness of a new investigational drug combination using alemtuzumab, belatacept, and sirolimus when given with or without donor bone marrow.

This combination of medicines has not been tested before in humans. Alemtuzumab (Campath) is approved for use in some types of white blood cell cancers, but is considered investigational in transplant patients. Belatacept is now FDA approved and is being studied in transplant patients. Sirolimus (Rapamune) is approved for use in transplant patients, but its use with belatacept and alemtuzumab is investigational.

In the initial 20 subjects enrolled in the study, half tested whether an infusion of bone marrow from the kidney donor would improve the effect of these drugs. This bone marrow infusion was also considered investigational.

Enrollment of 20 additional subjects began in January, 2013. The donor bone marrow infusion has been eliminated. Enrollment was open to primary living and deceased donor kidney recipients. Enrollment was closed as of 8/12/2014.

DETAILED DESCRIPTION:
This study will be a single-center, open-label,proof of concept study in non-human leukocyte antigen (HLA)-identical living and deceased donor renal transplants. The initial 20 subjects were randomized to either receive/not to receive a single donor bone marrow infusion in addition to the investigational combination of alemtuzumab, belatacept, and sirolimus. Since the bone marrow infusion has been eliminated in the second group of 20 subjects, no randomization was required. All recipients in the second group of 20 subjects will receive the same investigational combination of alemtuzumab, belatacept, and sirolimus.

At the time of transplant, participants will receive a 3-hour IV infusion of 30 mg. of alemtuzumab. Participants will receive a combination of sirolimus and belatacept for at least one year. At that time, eligible participants will consent to and begin oral immunosuppressive withdrawal or continue therapy through study close. Sirolimus will first be weaned by halving the dose and/or increasing the dosing interval over at least a 2-6 month period. After sirolimus is discontinued, participants will remain on monthly IV belatacept monotherapy indefinitely.

Follow-up will continue for at least five years. If subjects are successfully weaned from oral immunosuppression during their participation in this trial, no other alternative therapy will be warranted. Since belatacept is now FDA approved, subjects will be eligible to continue this therapy after their study participation has ended.

ELIGIBILITY:
Inclusion Criteria:

* Recipients age 18 or older of an HLA-non-identical, living or deceased donor kidney transplant.
* A willing renal donor who consents for subsequent donation of donor blood for testing throughout the follow-up period and for use of his/her kidney in this experimental study.

Exclusion Criteria:

* Immunosuppressive drug therapy within 1 year prior to enrollment.
* Active malignancy or history of malignancy within 5 years of enrollment.
* Any history of blood malignancy or lymphoma.
* Any known immunodeficiency syndrome, including HIV infection.
* Absence of Epstein-Barr virus (EBV) or cytomegalovirus (CMV) specific antibodies in cases with evidence of EBV and/or CMV infection.
* Women of child-bearing potential unwilling or unable to use an acceptable method of birth control.
* Women who are pregnant or breastfeeding at the time of enrollment or study drug administration.
* Donor age <18 years.
* Subjects with protocol-specific etiologies of underlying renal disease.
* Subjects with a positive T-cell lymphocytic crossmatch or historical evidence of donor specific alloantibody by solid phase or flow-based detection methods.
* Prior solid organ transplant or potential to require a concurrent organ or cell transplant.
* Positive Hepatitis B or C antibodies and polymerase chain reaction (PCR) positive for the same.
* Active tuberculosis (TB) requiring treatment within the previous 3 years.
* Known positive purified protein derivative (PPD) unless chest x-ray is negative or treatment for latent TB has been completed.
* Active infection or other contraindications.
* History of drug or alcohol abuse within the past 5 years.
* Psychotic disorders which would interfere with adequate study follow-up.
* Active peptic ulcer disease, chronic diarrhea, or gastric malabsorption.
* All women 40 years or older with first degree family history of breast cancer will be required to have a screening mammogram within 6 months of study enrollment.
* Subjects with suspicion of breast malignancy which cannot be ruled out will be excluded.
* Belatacept use within 30 days prior to the day 1 visit.
* Prisoners or individuals who are involuntarily incarcerated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-12; Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Guasch, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia

REFERENCES:
- [Background] Xu H, Mehta AK, Gao Q, Lee HJ, Ghali A, Guasch A, Kirk AD. B cell reconstitution following alemtuzumab induction under a belatacept-based maintenance regimen. Am J Transplant. 2020 Mar;20(3):653-662. doi: 10.1111/ajt.15639. Epub 2019 Nov 13. PMID 31596034
- [Result] Xu H, Bendersky VA, Brennan TV, Espinosa JR, Kirk AD. IL-7 receptor heterogeneity as a mechanism for repertoire change during postdepletional homeostatic proliferation and its relation to costimulation blockade-resistant rejection. Am J Transplant. 2018 Mar;18(3):720-730. doi: 10.1111/ajt.14589. Epub 2017 Dec 12. PMID 29136317
- [Result] Xu H, Samy KP, Guasch A, Mead SI, Ghali A, Mehta A, Stempora L, Kirk AD. Postdepletion Lymphocyte Reconstitution During Belatacept and Rapamycin Treatment in Kidney Transplant Recipients. Am J Transplant. 2016 Feb;16(2):550-64. doi: 10.1111/ajt.13469. Epub 2015 Oct 5. PMID 26436448
- [Result] Kirk AD, Guasch A, Xu H, Cheeseman J, Mead SI, Ghali A, Mehta AK, Wu D, Gebel H, Bray R, Horan J, Kean LS, Larsen CP, Pearson TC. Renal transplantation using belatacept without maintenance steroids or calcineurin inhibitors. Am J Transplant. 2014 May;14(5):1142-51. doi: 10.1111/ajt.12712. Epub 2014 Mar 31. PMID 24684552
- [Derived] Xu H, Lee HJ, Schmitz R, Shaw BI, Li S, Kirk AD. Age-related effects on thymic output and homeostatic T cell expansion following depletional induction in renal transplant recipients. Am J Transplant. 2021 Sep;21(9):3163-3174. doi: 10.1111/ajt.16625. Epub 2021 May 20. PMID 33942491

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in December 2007 and all study activities completed on July 1, 2017 Participants were enrolled from patients of Emory University Hospital and the Emory Clinic in Atlanta, Georgia.
Groups:
- Immunosuppresive Medication Combination: Renal transplant recipients receiving an experimental combination of immunosuppressive medications. Participants received a single dose of alemtuzumab on the day of transplantation and receive belatacept and sirolimus for one year.
Period: Overall Study
Arm/Group | Immunosuppresive Medication Combination
Started | 40
Completed | 38
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Immunosuppresive Medication Combination
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 46.5 [20 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40
Also received a bone marrow transfusion [Count of Participants; unit: Participants] | 9
Type of Transplant [Count of Participants; unit: Participants]
  Living donor transplant | 30
  Deceased donor transplant | 10
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 26.0 [18.6 to 37.3]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Successfully Withdrawn From Oral Immunosuppression
Description: The primary endpoint is the number of patients successfully withdrawn from oral immunosuppression (sirolimus) for one year after their last dose of sirolimus. After taking sirolimus for one year, participants meeting certain pre-specified criteria were offered the opportunity to wean from sirolimus and continue with belatacept monotherapy. To be eligible for weaning of sirolimus, participants were required to have a kidney biopsy negative for all signs of rejection, including borderline findings.
Time Frame: Year 2
Population: This analysis includes participants meeting criteria to wean from sirolimus who also opted to attempt sirolimus weaning.
Measure: Count of Participants; unit: Participants
Arm/Group | Immunosuppresive Medication Combination
Number analyzed (Participants) | 19
Participants
  Successful weaning | 12
  Failed weaning | 7

2. Secondary Outcome: Number of Participants Experiencing Costimulation Blockade-resistant Rejection (CoBRR)
Description: Assessment of the proposed therapies to prevent biopsy proven acute rejection, also known as CoBRR, was determined by the number of participants experiencing CoBRR at 1, 3 and 5 years post-transplant.
Time Frame: Year 1, Year 3, Year 5
Population: Between the 3 and 5 year assessments, one participant was removed for no longer meeting eligibility criteria and one participant withdrew from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Immunosuppresive Medication Combination
Number analyzed (Participants) | 40
Participants
  Year 1 | 0
  Year 3 | 0
  Year 5: number analyzed (Participants) | 38
  Year 5 | 0

3. Secondary Outcome: Number of Participants Experiencing Chronic Allograft Nephropathy (CAN)
Description: Assessment of biopsy proven chronic allograft nephropathy at 1, 3 and 5 years post-transplant is presented as the number of participants experiencing CAN.
Time Frame: Year 1, Year 3, Year 5
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Immunosuppresive Medication Combination
Number analyzed (Participants) | 40
Participants
  Year 1 | 0
  Year 3 | 0
  Year 5: number analyzed (Participants) | 38
  Year 5 | 0

4. Secondary Outcome: Number of Participants With BK Viremia
Description: The number of participants experiencing BK viremia, an opportunistic infection, during the study is presented here.
Time Frame: Up to Year 5
Measure: Count of Participants; unit: Participants
Arm/Group | Immunosuppresive Medication Combination
Number analyzed (Participants) | 40
Participants | 17

5. Secondary Outcome: Number of Participants Developing Donor-specific Alloantibody (DSA)
Description: Long term assessment of donor-specific immune responsiveness after prolonged therapy with belatacept (with or without sirolimus), and during and following drug withdrawal as determined by in vitro alloresponsiveness in carboxyfluorescein succinimidyl ester (CFSE) mixed lymphocyte reactivity and intracellular cytokine staining (ICCS).
Time Frame: Up to Year 5
Measure: Count of Participants; unit: Participants
Arm/Group | Immunosuppresive Medication Combination
Number analyzed (Participants) | 40
Participants | 5

6. Secondary Outcome: Number of Participants With Surviving Grafts
Description: The number of participants whose grafts survived without graft failure at each follow up time point is presented here.
Time Frame: Year 1, Year 3, Year 5
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Immunosuppresive Medication Combination
Number analyzed (Participants) | 40
Participants
  Year 1 | 40
  Year 3 | 40
  Year 5: number analyzed (Participants) | 38
  Year 5 | 36

7. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: Graft function was assessed throughout the study by the estimated glomerular filtration rate. The eGFR indicates the percentage of kidney function that a person has based on creatinine, age, body size, and gender. An eGFR of below 60 indicates chronic kidney disease. A higher eGFR means that there is greater kidney function.
Time Frame: Year 1, Year 3, Year 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Immunosuppresive Medication Combination
Number analyzed (Participants) | 40
mL/min/1.73m^2
  Year 1 | 70 (23)
  Year 3 | 67 (21)
  Year 5: number analyzed (Participants) | 38
  Year 5 | 71 (19)

ADVERSE EVENTS:
Time Frame: Information on adverse events were collected from the time of initiation of the investigational product through the 5 year follow up visit.
Description: Only adverse events that were related to the study medications (Alemtuzumab, Sirolimus, Belatacept) were recorded during the course of this study. Certain adverse events that occur commonly in this study population were not recorded as an adverse event, unless it was believed to be associated with the study medications or met the definition of a serious adverse event. Pre-existing conditions were not considered adverse events.
Arm/Group | Immunosuppresive Medication Combination
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 14/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immunosuppresive Medication Combination (N=40)
Shingles (Skin and subcutaneous tissue disorders) | 2
HHV-8/Kaposi's sarcoma (Skin and subcutaneous tissue disorders) | 1
Incisional hernia (Surgical and medical procedures) | 2
Mouth ulcers (sirolimus-associated) (Skin and subcutaneous tissue disorders) | 9
Pericardial effusion (Cardiac disorders) | 1
Edema (General disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT00565773/Prot_SAP_000.pdf